CLINICAL TRIAL: NCT07272434
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy, Immunogenicity, and Safety of a Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell) in Adults Aged 60 Aears and Above
Brief Title: Phase III Clinical Trial of the Recombinant Respiratory Syncytial Virus Vaccine ( CHO Cell)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government); Hunan Provincial Center for Disease Control and Prevention (Other); Hubei Provincial Center for Disease Control and Prevention (Other); Shaanxi Provincial Center for Disease Control and Prevention (Other); Guangdong Center for Disease Prevention and Control (Other Government); Shandong Province Centers for Disease Control and Prevention (Other); Sichuan Center for Disease Control and Prevention (Other Government); Hebei CDC ,China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-900-002
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Group (Experimental): Participants will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell)
- Placebo Group (Placebo Comparator): Participants will receive single dose of placebo, by IM injection into the deltoid region of the arm.
  Interventions: Biological: Placebo (Saline solution)

INTERVENTIONS:
Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell) — 0.5 mL per dose
  Arms: Vaccine Group
Biological: Placebo (Saline solution) — 0.5 mL per dose
  Arms: Placebo Group

SUMMARY:
This study will evaluate the efficacy of the Recombinant RSV vaccine(CHO cell) vaccine in preventing lower respiratory tract diseases(LRTD) caused by RSV in adults≥ 60 years of following a single dose of the RSV vaccine(CHO cell) vaccine .This study will also assess if the vaccine is safe and induces an immune response.

DETAILED DESCRIPTION:
A total of 25000 adults aged 60 years and above will be enrolled, stratified into 60-69 and ≥70 years of age. All Participants will randomly receive investigational vaccine or placebo at a ratio of 1:1. Efficacy and safety will be assessed in all Participants, while immunogenicity will be assessed in a subset of 1200 Participants in a selected trial site.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female can provide legal identification at the time of enrollment, and is 60 years of age or older (women are required to be infertile).

   (Note: Women with infertility include those who have been menopausal or have undergone sterilization (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy, etc.)
2. Be able to understand the trial procedures, risks and benefits and voluntarily agree to participate in the study and sign an informed consent.
3. Be able to participate in all scheduled visits and comply with the protocol requirements
4. Participants with stable health conditions considered by the investigator. Stable health conditions refer to patients with chronic diseases whose conditions are stable (regardless of whether they have received specific treatment or not), such as diabetes, hypertension, chronic obstructive pulmonary disease, asthma, etc. If the researcher determines that the condition is stable, they may be allowed to participate in this trial.

Exclusion Criteria:

Participants who meet any of the following exclusion criteria will not be allowed to enter the study (if the number of participants is not yet met, if the criteria described in "*" are met during screening, repeated screening may be performed)

1. *Axillary temperature>37.3℃.
2. History of RSV infection within 6 months before enrollment.
3. *New onsets of respiratory tract infection symptoms like cough, sputum, shortness of breath, wheezing, fever, runny nose or nasal congestion within 7 days before enrollment.
4. *Acute diseases or acute exacerbation of chronic disease within 3 days before vaccination.
5. *Within 3 days before enrollment, antipyretic and analgesic drugs (except enteric-coated aspirin tablets for the prevention of cardiovascular and cerebrovascular diseases) and antihistamines were used
6. Those who are allergic to the known components in the test vaccine [saponin (QS-21), dioleoyl phosphatidylcholine (DOPC), cholesterol, sucrose, sodium dihydrogen phosphate, anhydrous sodium dihydrogen phosphate, polysorbate 80, sodium chloride, hydrochloric acid and sodium hydroxide] Those who have a history of severe allergies after any vaccination or medication use [such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), severe urticaria, etc.] or serious adverse reactions.
7. Asplenia or functional asplenia, and any condition leading to asplenia or splenectomy.
8. Those who have had or are currently suffering from malignant tumors (except for clinically cured carcinoma in situ and papillary thyroid carcinoma).
9. Patients are diagnosed with autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease and autoimmune thyroid disease.
10. Persons with known or suspected immunodeficiency disorders [e.g. primary or secondary immunodeficiency, or diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus infection or immunosuppressive/cytotoxic agent therapy (e.g. cancer chemotherapy, organ transplantation or autoimmune disease treatment) resulting in confirmed or suspected immunosuppression or immunodeficiency].
11. According to the investigator's assessment,there is any disease that may make intramuscular injections unsafe, such as a history of thrombocytopenia or other coagulation disorders.
12. Those who have a history or are currently suffering from severe clinical diseases that have not been cured (such as severe cardiovascular and cerebrovascular diseases, liver and kidney diseases, respiratory system diseases, diabetes with complications, major surgeries, etc.) and may affect the evaluation of the trial.
13. Those who have had or are currently suffering from thrombotic diseases.
14. Patients with a history of untreated TB or active TB at enrollment.
15. *Hypertension with poor medication control (on-site blood pressure measurement before vaccination: systolic blood pressure≥150mmHg and/or diastolic blood pressure≥100mmHg).
16. Those with severe arrhythmias (such as atrial fibrillation).
17. Those with a history or family history of convulsions, epilepsy, congenital brain hypoplasia, mental illness, etc., or a history of brain nerve tissue damage caused by other serious neurological diseases (such as brain tumors, cerebral hemorrhage, brain infections, chemical drug poisoning, etc.).
18. Use of any experimental or unapproved product (drug, vaccine or medical device) other than the vaccine used in this trial or participate in other clinical trials within 30 days prior to enrollment or during the trial period.
19. *Within 14 days prior to enrollment, any non-live vaccine has been administered, or within 28 days, a live vaccine or nucleic acid vaccine has been administered.
20. Has received the RSV vaccine before.
21. Use of immunoglobulin and/or any blood preparation or plasma derivative, such as gamma globulin or intravenous human immunoglobulin, within 3 months prior to enrollment or plan to use during the trial
22. Within the 3 months prior to enrollment or if it is expected to be used for a long period during the trial (continuous for more than 14 days), immunosuppressive agents or other immunomodulatory drugs (such as long-term use of systemic glucocorticoids for ≥ 14 days, with a dose of ≥ 20mg/day prednisone or equivalent prednisone dose; local medications are allowed, such as ointments, eye drops, inhalants or nasal sprays, but the local medication dosage must not exceed the recommended dosage in the instructions)
23. Long-acting immunomodulatory drugs (such as infliximab) were used within 6 months before enrollment or during the planned trial period.
24. The researchers determined that the drinking behavior and/or drug abuse history that might affect the assessment of the trial (Note: within the last three months, men had an average of more than 14 standard drinks per week, and women had an average of more than 7 standard drinks per week; 1 standard drink contained 14g of alcohol, such as 360mL of beer or 45mL of 40% alcohol spirit or 150ml of wine.) Drug abuse refers to the repeated and excessive use of drugs with dependent characteristics or potential for dependence, which is not related to recognized medical needs and falls under non-medical purpose drug use.
25. Planned move to a location that will prohibit participating in the trial until study end;
26. Any condition that, in the opinion of the investigator, may affect the safety of the participant or the evaluation of the study results.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25000 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The first-time incidence rate per person-year of Lower Respiratory Tract Disease (LRTD). | From 14 days after vaccination until the end of the first RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by Reverse Transcription-Polymerase Chain Reaction（RT-PCR）.

SECONDARY OUTCOMES:
The first-time incidence rate per person-year of Acute Respiratory Illness (ARI). | From 14 days after vaccination until the end of the first RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of Severe Lower Respiratory Tract Disease (sLRTD). | From 14 days after vaccination until the end of the first RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of LRTD. | After vaccination, during the second RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of ARI. | After vaccination, during the second RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of sLRTD. | After vaccination, during the second RSV epidemic season,assessed up to 12 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of LRTD. | From 14 days after vaccination until the end of the second RSV epidemic season,assessed up to 24 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of ARI. | From 14 days after vaccination until the end of the second RSV epidemic season,assessed up to 24 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
The first-time incidence rate per person-year of sLRTD. | From 14 days after vaccination until the end of the second RSV epidemic season,assessed up to 24 months.
  A case caused by RSV-A and/or RSV-B as confirmed by RT-PCR.
Geometric Mean Titers (GMT) of Neutralizing Antibody against RSV-serotype A and RSV-serotype B. | At 14 days,1,12,24 and 36 months after vaccination
  Measured by Virus Neutralization Test.
Geometric Mean Fold Rise (GMFR) of Neutralizing Antibody against RSV-serotype A and RSV-serotype B | At 14 days,1,12,24 and 36 months after vaccination
  Measured by Virus Neutralization Test.
Geometric Mean Concentrations (GMC) of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | At 14 days,1,12,24 and 36 months after vaccination
  Measured by ELISA.
GMFR of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | At 14 days,1,12,24 and 36 months after vaccination
  Measured by ELISA.
Incidence, Intensity and Causality of adverse events(AEs) | Within 30 days after vaccination
  An AE includes any untoward medical occurrence in a patient or clinical investigation participants administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Incidence, Intensity and Causality of solicited AEs | Within 7 days after vaccination
  Solicited AEs include solicited local and general symptoms; Assessed solicited local AEs at injection site are pain, erythema, swelling, induration and itching; Assessed solicited general symptoms include fever, fatigue, headache, myalgia, nausea, vomiting, diarrhea, arthralgia and hypersensitivity.
Incidence, Intensity and Causality of unsolicited AEs | Within 30 days after vaccination
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation participants temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Incidence and Causality of Severe adverse events(SAEs) | Up to 12 months post vaccination
  SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in persistent or significant disability/incapacity or are congenital anomaly/birth defect.
Incidence and Causality of Adverse event of special interest (AESI) | Up to 12 months post vaccination
  Adverse events of special interest include potential immune-mediated diseases and atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (8):
- China (8):
  - Guangdong Provincial Center for Disease Control and Prevention, Guangzhou, Guangdong
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Henan Center for Disease Control and Prevention, Zhengzhou, Henan
  - Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei
  - Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan
  - Shaanxi Provincial Center for Disease Control and Prevention, Xi'an, Shaanxi
  - Shandong Province Centers for Disease Control and Prevention, Jinan, Shandong
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No